CLINICAL TRIAL: NCT01503437
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-sequence, Two-period, Single-dose, Crossover Bioequivalence Study of Olanzapine 5 mg OD Tablets With Zyprexa Zydis 5 mg Tablets in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Olanzapine Orally Disintegrating Tablets, 5 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BE-170-OLAN-2006
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olanzapine OD Tablets 5 mg (Experimental): Olanzapine OD Tablets 5 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Olanzapine OD Tablets 5 mg
- Zyprexa Zydis 5 mg Tablets (Active Comparator): Zyprexa Zydis 5 mg Tablets of Cardinal Health, UK
  Interventions: Drug: Olanzapine OD Tablets 5 mg

INTERVENTIONS:
Drug: Olanzapine OD Tablets 5 mg — Olanzapine OD Tablets 5 mg of Dr. Reddy's Laboratories Limited
  Other Names: Zyprexa Zydis

SUMMARY:
The purpose of this study is to compare the single oral dose bioequivalence of olanzapine 5 mg OD tablets with Zyprexa Zydis 5 mg tablets under fasting conditions and to monitor adverse events and ensure safety of subjects.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two treatment, two-sequence, two-period, single-dose, crossover comparative bioequivalence study of Olanzapine 5 mg OD Tablets, of Dr. Reddy's Laboratories Limited and Zyprexa Zydis 5 mg Tablets of Cardinal Health in healthy, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human subjects within the age range of 18 to 45 years
* Non-smokers since at least six months
* Willingness to provide written informed consent to participate in the study
* Body-mass index of ≥18.5 kg/m2 and ≤ 24.9 kg/m2, with body weight not less than 50 kg
* Absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluations, medical history or physical examination during the screening
* Normal 12-lead ECG or one with abnormality considered to be clinically insignificant
* Normal chest X-ray PA view
* Comprehension of the nature and purpose of the study and compliance with the requirement of the protocol
* Female Subjects

  * of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams. Jellies, diaphragm, intrauterine device (IUD), or abstinence, or
  * postmenopausal for at least 1 year, or
  * surgically sterile (bilateral tubal ligation. bilateral oophorectomy, or hysterectomy has been performed on the subject

Exclusion Criteria:

* Personal / family history of allergy or hypersensitivity to olanzapine or allied drugs
* Past history of anaphylaxis or angioedema
* Any major illness in the past three months or any clinically significant ongoing chronic medical illness e.g. congestive heart failure, hepatitis, pancreatitis etc.
* Presence of any clinically significant abnormal values during screening e.g. significant abnormality of liver Function Test (LFT), Renal (kidney) Function Test (RFT), etc.
* Any cardiac, renal or liver impairment, any other organ or system impairment
* History of seizure or psychiatric disorders
* Presence of disease markers of HIV 1 and 2, and hepatitis Band C virus
* Consumption of alcohol for more than two years, or consumption of more than three alcoholic drinks per day or consumption of alcohol within 48 hours prior to dosing and during the study [one drink is equal to one unit of alcohol [ one glass Wine, half plnt boor, and one measure (one ounce) of spirit).
* Consumption of xanthine containing derivatives (coffee, tea, cola drinks. chocolate) within 48 hours before check-in of each period
* Use of any recreational drug or a history of drug addiction
* Participation in any clinical trial within the past 3 months
* Inaccessibility of veins in left and right arm
* Donation of blood (one unit or 350 mL) within 3 months prior to receiving the first dose of study medication
* Receipt of any prescription drug therapy within four weeks or over-the-counter (OTC) drugs within two weeks prior to receiving the first dose of study medication or repeated use of drugs Within the last four weeks
* An unusual diet, for whatever reason e.g. low sodium diet, for two weeks prior to receiving any medication and through out subject's participation in the study
* Consumption of grapefruit- containing food or beverages within 7 days prior to receiving the first dose of study medication in both the periods
* Recent history of dehydration from diarrhea, vomiting or any other reason within a period of 24 hours prior to the study
* Female volunteers demonstrating a positive pregnancy screen or currently breast-feeding
* Having an occupation or requirement of driving a vehicle or operate a complex machinery before 21 days of taking the drug in both periods

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2006-11; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ghanashyam Rao, MBBS, Principal Investigator — Wellquest Clinical Research
Locations (1):
- Wellquest Clinical Research, Mumbai, Maharashtra, India